CLINICAL TRIAL: NCT05719324
Title: Checkpoint Inhibitors in Patients With Solid Tumors: a Retrospective Real-world Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-SR-219
Record Dates: First submitted 2023-01-31; First posted 2023-02-08 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Immunotherapy
Keywords: Immunotherapy; Checkpoint inhibitor; Solid tumor; Predictor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective clinical study aimed at observing and evaluating the effectiveness and safety of checkpoint inhibitors in the treatment of patients with solid tumors in actual clinical applications. To explore predictors of efficacy patients with unresectable solid tumors receiving checkpoint inhibitors and develop and further validate predictive models.

DETAILED DESCRIPTION:
The clinical data of patients with unresectable solid tumors were collected retrospectively, who received two or more cycles of checkpoint inhibitor therapy. The progression-free survival (PFS), overall survival (OS) and related adverse reactions of the patients were followed up. To screen prognostic factors, develop predictive models and visualize them as nomograms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old and gender is not limited.
* Patients with unresectable solid tumors confirmed by pathology or histology.
* Patients received checkpoint inhibitor therapy for 2 cycles or more.

Exclusion Criteria:

* Have a history of immunodeficiency, or suffer from other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation.
* Pre-existing thyroid dysfunction that cannot be maintained within the normal range even with medical treatment.
* Pregnant or breastfeeding women.
* Those who have a history of psychotropic drug abuse and cannot quit or have mental disorders.
* The investigator judges that other conditions are not suitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable solid tumors confirmed by histopathology or cytology, and continuously treated with checkpoint inhibitor based treatment for 2 cycles or more.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS） | Up to 24 months.
  PFS is defined as the time from initiation of checkpoint inhibitors until disease progression or death, whichever comes first.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 24 months.
  OS is defined as the time from initiation of checkpoint inhibitors to death or last follow-up.

OTHER OUTCOMES:
Objective response rate (ORR) | Up to 24 months.
  ORR is defined as the percentage of patients achieving complete response and partial response.
Disease Control Rate (DCR) | Up to 24 months.
  DCR is defined as the percentage of patients achieving complete response, partial response and stable disease.
Adverse events (AE) | Up to 24 months.
  AE includes abnormalities in clinical symptoms, vital signs and laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: Lingxiang Liu, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China